CLINICAL TRIAL: NCT00075023
Title: Evaluation of Efficacy and Mechanisms of Topical Thalidomide for Chronic Graft-Versus-Host-Disease Related Stomatitis
Brief Title: Effectiveness of Topical Thalidomide to Treat Chronic Graft-Versus-Host-Disease Related Stomatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unable to enroll adequate subjects
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Collaborators: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 040069; 04-NR-0069
Record Dates: First submitted 2003-12-30; First posted 2003-12-31 (Estimated); Results first posted 2015-11-04 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: Graft-versus-Host Disease; Stomatitis
Keywords: Stomatitis; Oropharyngeal pain; TNF-alpha; Allogeneic hematopoietic stem cell transplant; Inflammation; Thalidomide; Oral chronic graft-versus-host disease
MeSH Terms: conditions — Graft vs Host Disease; Stomatitis; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thalidomide gel (Experimental): Thalidomide gel 20 mg applied topically 4 times daily for 4 weeks to a maximum of 3 target oral ulcers
  Interventions: Drug: Thalidomide Gel
- Placebo (Experimental): Placebo gel with no Thalidomide applied topically 4 times daily for 4 weeks to a maximum of 3 target oral ulcers
  Interventions: Drug: Placebo Gel

INTERVENTIONS:
Drug: Thalidomide Gel
  Arms: Thalidomide gel
Drug: Placebo Gel
  Arms: Placebo

SUMMARY:
This study was designed to be conducted in 2 parts. The first part is a pilot study to test the effects of topical thalidomide gel 20mg applied to up to 3 oral ulcers in patients who have developed oral chronic graft-versus-host-disease (cGVHD)-related ulcerative stomatitis following allogeneic bone marrow/peripheral blood stem cell transplant (HSCT). Chronic GVHD may be related to increased levels of a cytokine called TNF-alpha (TNFa) following HSCT. Thalidomide's anti-inflammatory effects may lower TNFa levels, lead to healing of these oral ulcers, and decrease oral pain.

If the pilot study is successful, the second part of the study will be done. This will test the effects of a 0.1% (20mg) thalidomide mouthwash in treating oral cGVHD-related stomatitis in patients following allogeneic HSCT. Applying thalidomide directly to the GVHD-related mouth ulcer in gel form or to the entire oral cavity in mouthwash form rather than taking it in pill form may reduce the amount of drug that enters the blood stream and cause less side effects.

In the pilot study, participants will be randomly assigned to receive thalidomide gel 20mg or placebo (identical gel with no thalidomide) to use 4 times a day for 4 weeks. In the mouthwash study, participants will be randomly assigned to receive 0.1% 20mg thalidomide mouthwash or placebo (identical mouth rinse with no thalidomide) to use 4 times a day for 4 weeks. Participants will undergo the following procedures before beginning experimental treatment, then once a week for 4 weeks, and then approximately 8 weeks after the first visit:

* Interview about current medications and use of alcohol and cigarettes
* Self-report of mouth and throat pain
* Oral examination for stomatitis rating, and oral ulcer(s) measurement
* Quality of life questionnaire (repeated only at week 8 of the study)
* Mouth photography to measure and record the oral ulcer response to treatment
* Saliva sampling to look for proinflammatory cytokines (small proteins), including TNFa
* Oral ulcer exudate collected by filter paper to obtain fluid for measuring TNFa levels
* Gentle swabbing of oral ulcers to culture for virus, fungus, and bacteria that may be present
* Small punch biopsy of the area near the ulcer or affected area to check for presence of TNFa (repeated only at week 4 of the study)
* Blood sampling to monitor TNFa levels
* A urine pregnancy test for women who are able to have children (repeated at weeks 2, 4, and 8)

DETAILED DESCRIPTION:
Oncology patients undergoing allogeneic bone marrow/peripheral blood stem cell transplant (HSCT) frequently experience an allo-immune condition termed graft-versus-host-disease (GVHD). The pathogenesis of GVHD derives from an immune attack mediated by donor T-cells recognizing antigens expressed on normal tissues of the patient. This condition occurs in HSCT rather than autologous BMT because of disparities in minor histocompatibility antigens between donor and recipient, inherited independently of HLA genes (Lazarus, Vogelsang, and Rowe, 1997). GVHD may be conceptualized as a cytokine storm stemming from an outpouring of endogenous cytokines resulting in many tissue effects (Lazrarus et al, 1997). Oral chronic GVHD (cGVHD) presents with tissue atrophy and erythema, lichenoid changes (hyperkeratotic striae, patches, plaques, and papules) and pseudomembranous ulcerations typically occurring on the buccal and labial mucosa and the lateral tongue, mucoceles due to inflammation of minor salivary glands, and xerostomia (Lloid, 1995). The ulcerative phase often leads to a cascade of negative sequelae including oropharyngeal pain, critical treatment alterations or cessation, diminished capacity for food intake, and decreased quality of life.

Optimal treatment strategies for cGVHD-related ulcerative stomatitis and related oropharyngeal pain have not been established. Therefore, there is a critical need to examine the pathogenesis of and to evaluate interventions for cGVHD-related ulcerative stomatitis and related acute oropharyngeal pain in the randomized controlled clinical trial setting to both advance the science of cancer treatment-related oral complications and to improve patient care. We hypothesize that the mechanisms of tissue injury occurring at the mucosal level leading to cGVHD-related stomatitis are similar to other types of stomatitis, such as cancer chemotherapy-related stomatitis and aphthous stomatitis, and are therefore amenable to treatment with anti-inflammatory strategies. Therefore, the purpose of this study is to elucidate the role of inflammation in GVHD-related ulcerative stomatitis by testing the efficacy of a topical thalidomide gel on the resolution of cGVHD-related stomatitis and related oropharyngeal pain. The actions of thalidomide, which include inhibition of the release of tumor necrosis factor-alpha (TNFa) and resultant alteration of the inflammatory cascade, may provide insight into the role of local mucosal inflammation in cGVHD-related stomatitis.

This study will be conducted in two parts. The first part is a pilot study testing the effects of a thalidomide gel 20mg in patients who have developed oral cGVHD-related ulcerative stomatitis following allogeneic bone marrow/peripheral blood stem cell transplant (HSCT). Stomatitis is an inflammation of the lining of the throat and mouth that may lead to ulcers and pain in the mouth and throat. GVHD - a condition in which the donor cells see patient's cells as foreign and mount an immune response to them - may be related to increased levels of a substance called TNF-alpha (TNFa) following HSCT. Thalidomide's anti-inflammatory effects may lower TNFa levels and decrease cGVHD-related stomatitis and oral pain in these patients.

If this pilot study is successful, then the second part of the study will be conducted. The second part of this study will test the effects of a 0.1% (20mg) thalidomide mouthwash in treating oral cGVHD-related stomatitis in patients following allogeneic HSCT. Applying thalidomide directly to the GVHD-related mouth ulcer in gel form or to the entire oral cavity in mouthwash form rather than taking the thalidomide in pill form may reduce the amount of drug that enters the blood stream and cause fewer side effects.

Patients between 18 and 80 years of age who have received a HSCT and developed oral cGVHD-related stomatitis as confirmed by surgical biopsy may be eligible for this study. The only eligible female participants for the pilot study will be women who are unable to have children. In the pilot study, participants will be randomly assigned to receive thalidomide gel 20mg or placebo (a gel with no thalidomide) to use four times a day for 4 weeks. In the mouthwash study, participants will be randomly assigned to receive 0.1% 20mg thalidomide mouthwash or placebo (a mouth rinse with no thalidomide) to use four times a day for 4 weeks.

Participants will have the following data collected and undergo the following procedures before beginning experimental treatment, then once a week for 4 weeks, and then approximately 8 weeks after the first visit.

* Interview about current medications and use of alcohol and cigarettes.
* Self-report of mouth and throat pain ratings.
* Oral examination for stomatitis rating
* Quality of life questionnaire (The questionnaire is repeated only at week 8 of the study.).
* Mouth photography to measure and record the oral ulcer response to treatment.
* Saliva sampling to look for proinflammatory cytokines (small proteins), including TNFa.
* Oral ulcer exudate collected by filter paper to obtain fluid for measuring TNFa levels.
* Gentle swabbing of oral ulcers to culture for virus, fungus, and bacteria that may be present.
* Small punch biopsy of the area near the ulcer or affected area to check for presence of TNFa. (The punch biopsy is repeated only at week 4 of the study.)
* Blood sampling to monitor TNFa levels.
* A urine pregnancy test for women who are able to have children. (The pregnancy test is repeated at weeks 2, 4, and 8.)

ELIGIBILITY:
* INCLUSION CRITERIA:

Participating in HSCT or cGVHD protocols and willing to participate in this study concurrently;

Diagnosed with oral cGVHD stomatitis confirmed by surgical biopsy results;

Oral ulceration present

Able to understand and sign protocol informed consent;

Ages 18 to 80 years of age.

EXCLUSION CRITERIA:

Pregnant or lactating females;

For the proof of concept study, females who are not surgically sterilized by means of hysterectomy or tubal ligation;

For the main study, females of childbearing potential who do not agree to the use of two forms of highly effective contraception for at least four weeks prior, during, and for four weeks following the last dose of study drug;

Sexually active males who do not agree to the use of a latex condom while receiving study drug and for four weeks following the last dose of study drug;

Unwilling to follow precautions for use of thalidomide;

Unable to demonstrate appropriate use of study medication;

Concurrent use of non-protocol-related medications confounding assessment of the inflammatory response (antihistamines, non-steroidal anti-inflammatory drugs);

Allergic reaction to thalidomide;

Pre-existing oral infection, which might maximize the possibility of an infection or sepsis contributing to a drug-related adverse event;

Unwilling or unable to forego concurrent treatment for mucosal lesions and/or related oral pain (including topical steroids, viscous lidocaine, topical anti-fungals);

Requiring addition of new systemic therapy including thalidomide, steroids, or radiation therapy;

Use of sedatives (including CNS depressants);

Absolute neutrophil count (ANC) less than 750/mm(3)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2003-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Fall-Dickson, RN, PhD, Principal Investigator — NIH/NINR
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Background] Albandar JM, Brunelle JA, Kingman A. Destructive periodontal disease in adults 30 years of age and older in the United States, 1988-1994. J Periodontol. 1999 Jan;70(1):13-29. doi: 10.1902/jop.1999.70.1.13. PMID 10052767
- [Background] Antin JH, Ferrara JL. Cytokine dysregulation and acute graft-versus-host disease. Blood. 1992 Dec 15;80(12):2964-8. PMID 1467511
- [Background] Aucott DM, Ashley FP. Assessment of the WHO partial recording approach in identification of individuals highly susceptible to periodontitis. Community Dent Oral Epidemiol. 1986 Jun;14(3):152-5. doi: 10.1111/j.1600-0528.1986.tb01521.x. PMID 3459612
- [Derived] St John L, Gordon SM, Childs R, Marquesen M, Pavletic SZ, Wu TX, Cozzarelli T, Schroeder E, Saria MG, Fall-Dickson JM. Topical thalidomide gel in oral chronic GVHD and role of in situ cytokine expression in monitoring biological activity. Bone Marrow Transplant. 2013 Apr;48(4):610-1. doi: 10.1038/bmt.2012.178. Epub 2012 Sep 24. No abstract available. PMID 23000649
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2004-NR-0069.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Thalidomide Gel: Thalidomide Gel
- Placebo: Placebo Gel
Period: Pilot Study
Arm/Group | Thalidomide Gel | Placebo
Started | 5 | 5
Completed | 3 | 3
Not Completed | 2 | 2
Not completed — Physician Decision | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Period: Part Two
Arm/Group | Thalidomide Gel | Placebo
Started | 0 (Study was terminated after the pilot study. No participants entered Part Two.) | 0 (Study was terminated after the pilot study. No participants entered Part Two.)
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The sample size for the proof of concept study was calculated by using the data for aphthous ulcer percentage healing (personal communication with investigator) with topical thalidomide gel at 0 mg and 20 mg. This gave a total sample size of 60 using an alpha level = .05, beta = -.20 and a 2-tailed test. Assuming drop out rate of 10%, total is 66.
Groups:
- Total: Total of all reporting groups
Arm/Group | Thalidomide Gel | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Customized [Number; unit: participants]
  27-60 yrs | 5 | 5 | 10
Sex: Female, Male [Count of Participants; unit: Participants] — Total enrollment of 7 males and 3 females. Gender data not available for each arm.
  Participants
    Female | NA — Data not available per group | NA — Data not available per group | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | NA — Data not available per group | NA — Data not available per group | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage Change in Total Surface Area of Oral Ulceration.
Description: Mean percentage change in total surface area of oral ulceration
Time Frame: baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Thalidomide Gel | Placebo
Number analyzed (Participants) | 3 | 3
percentage change | -66 (NA) — Not available due to unavailable records | -59 (NA) — Not available due to unavailable records

ADVERSE EVENTS:
Groups:
- Adverse Events for All Participants: These are adverse events for participants as reported to the DSMB, without information related to treatment arm
Arm/Group | Thalidomide Gel | Placebo | Adverse Events for All Participants
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/0
Other Adverse Events (participants affected / at risk) | 2/5 | 2/5 | 6/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Thalidomide Gel (N=5) | Placebo (N=5) | Adverse Events for All Participants (N=10)
Increase in oral pain (General disorders) | 1 | 1 | 0/0 — Participant removed from study according to study stopping rules
Spouse pregnancy (Social circumstances) | 0 | 1 | 0/0 — Subject removed from study because he told research staff his wife was pregnant. He was removed due to concern over the risk of transmission of the study drug to the fetus.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0/0 — Subject hospitalized for non-protocol related penumonia and missed signficant doses of the study drug.
Dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0/0 | 1 — not related to drug
thrush (General disorders) | 0/0 | 0/0 | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0/0 | 2
Oral pain (General disorders) | 0/0 | 0/0 | 2
Sore throat (General disorders) | 0/0 | 0/0 | 2
headache (General disorders) | 0/0 | 0/0 | 1
tired (General disorders) | 0/0 | 0/0 | 1
peripheral neuropathy (General disorders) | 0/0 | 0/0 | 1
loss of appetite (Gastrointestinal disorders) | 0/0 | 0/0 | 1
somnolence (General disorders) | 0/0 | 0/0 | 1
rash (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 1

LIMITATIONS AND CAVEATS:
Small sample size due to difficult enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No